CLINICAL TRIAL: NCT05141643
Title: 18F-FAC PET Imaging to Quantify Gemcitabine Tumor Drug Uptake and Biodistribution in Pancreatic Cancer Patients
Brief Title: Imaging Study of 18F-FAC PET Scans to Assess Standard Treatment in People With Pancreatic Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-442
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer; pancreatic ductal adenocarcinoma; 18F-FAC; Memorial Sloan Kettering Cancer Center; 21-442
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with pancreatic ductal adenocarcinoma (PDAC) (Experimental): Participants will have histologically-confirmed pancreatic ductal adenocarcinoma (PDAC). The experimental design of this study is to perform a single [18F]-FAC PET scan prior to the administration of chemotherapy with an optional second [18F]-FAC PET scan procedure during SOC treatment to observe changes in tumor uptake and biodistribution. Patients will be offered a second [18F]-FAC PET scan procedure during their SOC treatment. This second scan will be optional.
  Interventions: Diagnostic Test: PET Scan

INTERVENTIONS:
Diagnostic Test: PET Scan — Participants will receive a minimum of 4 mCi (148 MBq) and up to a maximum of 10 mCi (370 MBq) of [18F]-FAC intravenously. Injection is performed in conjunction with a dynamic PET acquisition over a site of the disease (pre-selected based on the findings from a previous CT or MRI and FDG PET/CT study done for clinical purpose such as staging). Patients will be offered a second [18F]-FAC PET scan procedure during their SOC treatment. This second scan will be optional.
  Other Names: 18F-FAC PET Scan

SUMMARY:
The purpose of this study is to find out whether a pre-treatment PET scan using the experimental imaging tracer 18F-FAC can show how much of the standard chemotherapy for PDAC may be taken up by the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed (confirmed at MSKCC) PDAC
* Patients must be ≥ 18 years old
* Signed, written Institutional Review Board (IRB)-approved Informed Consent Form (ICF).
* Measurable or evaluable solid disease on computed tomography (CT) or magnetic resonance imaging (MRI) scan per RECIST v1.1.
* Karnofsky Performance Status ≥70%.
* Life expectancy ≥3 months.
* A negative serum pregnancy test, within 1 week of the procedure, if the patient is female of reproductive potential.

Exclusion Criteria:

* Patients who cannot undergo PET/CT scanning (i.e. because of weight limits, claustrophobia).
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Tumor drug uptake within PDAC tumors prior at pre-treatment baseline | Baseline
  The primary objective of this study is to obtain preliminary data of tumor drug uptake profile, concentration and distribution within PDAC tumors prior at pre-treatment baseline

SECONDARY OUTCOMES:
changes in [18F]-FAC drug uptake during or following SOC chemo- and/or radiation therapy. | 2 years
  To investigate changes in [18F]-FAC drug uptake and distribution during or following SOC chemo- and/or radiation therapy. Based on those patients who agree to undergo the second optional [18F]-FAC PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05141643/ICF_000.pdf